CLINICAL TRIAL: NCT07234682
Title: The Impact of the Anxiety-Sleep Disturbance Symptom Cluster on Cellular Immune Function and Quality of Life in Colorectal Cancer Patients During Chemotherapy: A Prospective Observational Study
Brief Title: Impact of Anxiety-Sleep Symptom Cluster on Immune Function and Quality of Life in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government)
Responsible Party: Principal Investigator, Xujin Guo, Principal investigator, Hebei Provincial Hospital of Traditional Chinese Medicine
Other Study IDs: HBZY2023-KY-050-01
Record Dates: First submitted 2025-09-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (MSI-H); Anxiety
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 5 mL peripheral blood sample was collected in an EDTA-containing tube for determination of absolute counts of T-lymphocyte subsets (CD3+, CD4+, CD8+) and natural killer (NK) cells.

GROUPS / COHORTS (2):
- Symptom Cluster Group (n=45): Patients with both clinically significant anxiety, defined as a Hospital Anxiety and Depression Scale - Anxiety (HADS-A) score of 8 or higher, AND significant sleep disturbance, defined as a Pittsburgh Sleep Quality Index (PSQI) global score greater than 5.
  Interventions: Other: standard-of-care chemotherapy
- No/Low Symptoms Group (n=58): Patients who do not meet the criteria for the Symptom Cluster group (i.e., do not have both clinically significant anxiety and significant sleep disturbance).
  Interventions: Other: standard-of-care chemotherapy

INTERVENTIONS:
Other: standard-of-care chemotherapy — This is an observational study where participants are categorized based on pre-existing symptoms (exposure), not assigned to an intervention by the investigator. Therefore, no formal "intervention" is being tested. The "Interventions" section as shown in the screenshot should be left blank. All participants received their standard-of-care chemotherapy as prescribed by their oncologist, which is the context of the study, not the intervention being evaluated.

SUMMARY:
This prospective observational study investigates the impact of the anxiety-sleep disturbance symptom cluster on cellular immune function and quality of life in colorectal cancer (CRC) patients undergoing chemotherapy. The study aims to determine if patients with clinically significant anxiety and sleep disturbance exhibit poorer immune cell profiles (e.g., T-cells, NK cells) and lower quality of life compared to patients with no or low symptoms.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) patients often experience debilitating symptom clusters during chemotherapy. The co-occurrence of anxiety and sleep disturbance is particularly common and may have a synergistic negative effect on patients' physiological and psychological well-being. This study was designed based on the principles of psychoneuroimmunology (PNI), which suggest that psychological states can influence the immune system. A total of 103 patients with Stage II-IV CRC undergoing standard chemotherapy were enrolled. Participants were assessed at the beginning of a chemotherapy cycle using validated questionnaires: the Hospital Anxiety and Depression Scale (HADS) for anxiety, the Pittsburgh Sleep Quality Index (PSQI) for sleep disturbance, and the EORTC QLQ-C30 for quality of life. Peripheral blood samples were collected to quantify lymphocyte subsets (CD3+, CD4+, CD8+, NK cells) via flow cytometry. Patients were stratified into a "Symptom Cluster" group (HADS-A ≥ 8 and PSQI > 5) and a "No/Low Symptoms" group. The study compares immune parameters and quality of life scores between the two groups and uses correlation and regression analyses to explore the relationships between symptom severity, immune function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Pathologically confirmed colorectal cancer (Stage II-IV);
3. Scheduled to receive a standard chemotherapy regimen (e.g., FOLFOX, FOLFIRI);
4. Able to understand and complete questionnaires.

Exclusion Criteria:

1. Severe cognitive impairment or psychiatric disorders other than anxiety/depression;
2. Concurrent use of psychotropic medications or sleep aids that could interfere with the study's primary measures;
3. Acute infection or autoimmune disease;
4. History of another primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of stage II-IV colorectal cancer undergoing a standard chemotherapy regimen (e.g., FOLFOX, FOLFIRI) at the Hebei Provincial Hospital of Traditional Chinese Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
CD4+ T-cell Count | Baseline
  Absolute count of helper T-cells (CD4+) in peripheral blood, measured by flow cytometry. Results are expressed as cells per microliter (cells/μL). A lower count indicates a more compromised immune status.
Global Health Status / Quality of Life Score | Baseline
  Assessed using the global health status/QoL scale from the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores are transformed to a 0-100 scale, with a higher score indicating a better global quality of life.

SECONDARY OUTCOMES:
CD3+ T-cell Count | Baseline
  Absolute count of total T-cells (CD3+) in peripheral blood, measured by flow cytometry and expressed as cells/μL.
CD8+ T-cell Count | Baseline
  Absolute count of cytotoxic T-cells (CD8+) in peripheral blood, measured by flow cytometry and expressed as cells/μL.
CD4+/CD8+ Ratio | Baseline
  The ratio of CD4+ T-cell count to CD8+ T-cell count, calculated from flow cytometry data. This ratio is an important marker of immune health.
Natural Killer (NK) Cell Count | Baseline
  Absolute count of Natural Killer (NK) cells in peripheral blood, measured by flow cytometry and expressed as cells/μL.
EORTC QLQ-C30 Functional Scales Scores | Baseline
  Scores from the five functional scales of the EORTC QLQ-C30: Physical, Role, Emotional, Cognitive, and Social Functioning. Scores range from 0 to 100, with higher scores indicating better functioning.
EORTC QLQ-C30 Symptom Scales Scores | Baseline
  Scores from the symptom scales of the EORTC QLQ-C30, including Fatigue, Pain, and Insomnia. Scores range from 0 to 100, with higher scores indicating a greater symptom burden.
Anxiety Severity Score | Baseline
  Assessed using the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). The scale consists of 7 items, with a total score ranging from 0 to 21. A score of ≥8 indicates clinically significant anxiety.
Sleep Disturbance Severity Score | Baseline
  Assessed using the global score of the Pittsburgh Sleep Quality Index (PSQI). The global score ranges from 0 to 21. A score >5 indicates significant sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei, China